CLINICAL TRIAL: NCT00148317
Title: A Sequential Phase II Trial of the Combination of Bortezomib (VELCADE), Dexamethasone (DECADRON) and Pegylated Liposomal Doxorubicin (DOXIL) Followed by High Dose Cyclophosphamide in Multiple Myeloma Patients
Brief Title: Phase II Study of Velcade, Decadron, and Doxil Followed by Cyclophosphamide in Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0504007841
Record Dates: First submitted 2005-09-02; First posted 2005-09-07 (Estimated); Results first posted 2017-07-18 (Actual); Last update posted 2017-07-18 (Actual); Status verified 2017-06

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; Dexamethasone; Calcium Dobesilate; liposomal doxorubicin; Cyclophosphamide; Filgrastim

STUDY DESIGN:
Intervention Model Description: Consolidation: All patients will receive 2 cycles of bortezomib (VEL) and dexamethasone (DEX). Patients who achieve a complete response after 2 cycles will receive 4 additional cycles of VEL/DEX before mobilization.
  Patients who do not achieve at least a partial response after 2 cycles will receive 4 more cycles of VEL/DEX plus DOXIL.
  Patients who achieve a partial response after 2 cycles on VEL/DEX, will continue this combination for 2 more cycles. Patients who achieve a complete response after 4 cycles will receive 2 additional cycles of VEL/DEX before mobilization. Patients who remain with a partial response after 4 cycles of VEL/DEX will receive 2 additional cycles of the combination of VEL/DEX plus DOXIL.
  Mobilization: Patients who complete 6 cycles of consolidation will proceed to mobilization. Patients will receive one cycle of VEL plus high dose CYTOXAN followed by G-CSF beginning 24 hours after CYTOXAN given for a total of 10 daily doses.

ARMS (1):
- Treatment Arm (Experimental)
  Interventions: Drug: Bortezomib; Drug: dexamethasone; Drug: liposomal doxorubicin; Drug: cyclophoshamide; Drug: filgrastim

INTERVENTIONS:
Drug: Bortezomib — During Induction Phase (6 cycles): Bortezomib 1.3 mg/m2 on days 1, 4, 8, and 11 During 21-day mobilization cycle (1 cycle): Bortezomib 1.3 mg/m2 on days 1, 4, 8, and 11
  Other Names: velcade
Drug: dexamethasone — During Induction Phase (6 cycles): dexamethasone 40 mg on days 1-4, 8-11, and 15-18
  Other Names: decadron
Drug: liposomal doxorubicin — If patients achieve less then a PR during the induction phase after 2 cycles, or less then a CR after 4 cycles: Liposomal doxorubicin was added at 30 mg/m2 on day 4 for the remaining cycles
Drug: cyclophoshamide — During the 21 day mobilization phase (1 cycle): cyclophosphamide at 3 g/m2 on day 8
  Other Names: cytoxan
Drug: filgrastim — During the 21 day mobilization phase (1 cycle): 10 μg/kg/day for 10 consecutive days starting 24 hours after cyclophosphamide administration on day 9
  Other Names: neupogen

SUMMARY:
PRIMARY STUDY OBJECTIVES

* To evaluate the efficacy of the combination of bortezomib, dexamethasone, with and without DOXIL, followed by high-dose cyclophosphamide as a therapy for two different subsets of multiple myeloma patients:

  1. Patients post first line therapy
  2. Patients with relapsed/refractory disease who are bortezomib-naïve
* To evaluate the safety of the combination of bortezomib and dexamethasone, with and without DOXIL, followed by high-dose cyclophosphamide as therapy for patients with multiple myeloma.

SECONDARY STUDY OBJECTIVES

* To evaluate the role of the combination of bortezomib dexamethasone, with and without DOXIL, followed by high-dose cyclophosphamide on the ability to collect > 10 x 106 CD34+ cells/kg in < 7 collections (for both subsets of multiple myeloma patients).
* To evaluate the survival of patients who receive the combination of bortezomib dexamethasone, with and without DOXIL, followed by high-dose cyclophosphamide (for both subsets of patients).

ELIGIBILITY:
Inclusion Criteria:

* Subject must voluntarily sign and understand written informed consent.
* Confirmed diagnosis of multiple myeloma as specified by the SWOG criteria and is detailed in Appendix I.
* Measurable disease as defined the following:

  1. For patients post induction therapy, any measurable paraprotein in the serum or urine and/or any plasmacytoma present on physical exam or imaging.
  2. For patients with relapsed/refractory disease, > 0.5 g/dL serum monoclonal protein, > 0.1 g/dL serum free light chains, > 0.2 g/24 hrs urinary M-protein excretion, and/or measurable plasmacytoma(s).
* Age > or = than 18 years at the time of signing the informed consent form.
* Karnofsky performance status> or =70% (>60% if due to bony involvement of myeloma).
* Group A (post-induction therapy)- patients who have received only one prior treatment regimen (eg VAD, Thal/Dex, BLT-D, MP, BiRD, or DVd) with at least 20 patients having received a Revlimid based regimen or Group B(>1st line of therapy)- patients with relapsed/refractory multiple myeloma who have received two or more prior treatment regimens .
* If the patient is a woman of childbearing age, she must have a negative serum or urine pregnancy test within 7 days of starting study and must use effective contraception throughout the course of the study.
* Life expectancy > 12 weeks.
* Absolute neutrophil count (ANC)> or = 1500 cells/mm3 (> or = 1000 for patients with bone marrow biopsy displaying > 50% involvement by myeloma)
* Platelets count > or = 50,000/mm3 (> or = 30,000 for patients with bone marrow biopsy displaying > 50% involvement by myeloma)
* Hemoglobin > 9.0 g/dL
* Serum SGOT/AST <3.0 x upper limits of normal (ULN)
* Serum SGPT/ALT <3.0 x upper limits of normal (ULN)
* Serum creatinine < 2.5 mg/dL or creatinine clearance > 40ml/min
* Serum total bilirubin < 1.5 x ULN
* Patients must have a MUGA scan with LVEF >50%

Exclusion Criteria:

* Patients with non-secretory MM (no measurable monoclonal protein, free light chains, and/or M-spike in blood or urine) unless measurable disease is available with imaging techniques such as MRI and PET scan.
* Prior treatment with bortezomib.
* Peripheral neuropathy of > Grade 2 as defined by CTCAE Version 3.0 (see Appendix II)
* History of allergic reactions to compounds containing mannitol, bortezomib, conventional formulation of doxorubicin HCL or the components of DOXIL.
* Prior history of other malignancies (except for basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix or breast) unless disease free for ³ 5 years.
* NYHA Class III or IV heart disease. History of active unstable angina, congestive heart disease, serious uncontrolled cardiac arrhythmia or myocardial infarction within 6 months.
* Female patients who are pregnant or breastfeeding. Women of childbearing potential and men must agree to use adequate contraception prior to study entry and for the duration of study participation.
* Known HIV or hepatitis A, B, or C positivity
* Active viral or bacterial infections or any coexisting medical problem that would significantly increase the risks of this treatment program.
* Any concurrent, uncontrolled medical condition, laboratory abnormality, or psychiatric illness which could place him/her at unacceptable risk, including, but not limited to, uncontrolled hypertension, uncontrolled diabetes, active uncontrolled infection, and/or acute chronic liver disease (i.e., hepatitis, cirrhosis).
* No prior anti-myeloma therapy within 2 weeks of treatment initiation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2005-06; Primary Completion 2011-02 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ruben Niesvizky, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Medical College of Cornell University, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Consolidation (VEL + DEX)
Arm/Group | Overall Study
Started | 38
DOXIL Added at Cycle 3 | 16
DOXIL Added at Cycle 5 | 12
no DOXIL Added | 10
Completed | 38
Not Completed | 0
Period: Mobilization (VEL+CYTOXAN+FILGRASTIM)
Arm/Group | Overall Study
Started | 38
Completed | 27
Not Completed | 11
Not completed — Adverse Event | 8
Not completed — Lack of Efficacy | 2
Not completed — unable to tolerate | 1

BASELINE CHARACTERISTICS:
Groups:
- Treatment Arm (All Patients): Bortezomib, Dexamethasone, Pegylated Liposomal Doxorubicin, Cyclophosphamide: Bortezomib 1.3 mg/m2 days 1, 4, 8, 11 (initial cycles) Dexamethasone 40 mg Days 1-4, 8-11, 15-18 (initial cycles) Doxil 30 mg/m2 Day 4 of subsequent cycles
Arm/Group | Treatment Arm (All Patients)
Number analyzed (Participants) | 38
Age, Continuous [Median (Full Range); unit: years] | 61 [27 to 76]
Age, Customized [Count of Participants; unit: Participants]
  Age <70 years | 34
  Age > or = 70 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 34
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 26
  More than one race | 0
  Unknown or Not Reported | 5
Beta-2 Microglubilin [Median (Full Range); unit: mg/L] | 2.05 [1.0 to 10.2]
Serum Albumin [Median (Full Range); unit: g/dL] | 3.5 [2.0 to 4.3]
Durie Salmon Staging System [Number; unit: participants] — The Durie Salmon Staging System was used to assess patients status. Stage 1A is associated with a better outcome & a low tumor burden, stage 2A with a intermediate outcome and tumor burden, and stage 3A with a worse outcome & higher tumor burden. Criteria for staging is based on multiple factors including hematology values, disease burden, and renal function. The staging system can be found here: https://www.themmrf.org/multiple-myeloma/prognosis/myeloma-stages/durie-salmon-staging-system/ As assessed by the treating physician, the 1a subject:had active myeloma based on the IMWG criteria.
  participants
    1a | 1
    2a | 19
    3a | 17
    3b | 1
International Staging System [Number; unit: participants] — Measure Description: Stage I ß2-M < 3.5 mg/dL and albumin =3.5 g/dL Stage II Neither stage I nor stage III Stage III ß2-M ≥ 5.5 mg/L
  participants
    I | 18
    II | 17
    III | 3
Abnormalities by FISH [Number; unit: participants] — Cytogenetic abnormalities were assessed in patients using fluorescence in situ hybridization (FISH), which detects chromosomal abnormalities. Del (17p), t(4;14), and t (14;16) were considered High Risk cytogenetic abnormalities. All other abnormalities were considered standard risk cytogenetics.
  participants
    trisomy 11 | 10
    hyperdiploidy | 7
    t (4;14) | 4
    p53 | 4
    del (17p) | 1
    t (11;14) | 5
    t (14;16) | 2
    none | 16
Prior induction therapy [Number; unit: participants]
  lenalidomide + dexamethasone ± BIAXIN | 21
  Thalidomide + lenalidomide + dexamethasone± BIAXIN | 8
  Thalidomide + dexamethasone | 3
  thalidomide only | 2
  pulsed dexamethasone only | 2
  melphalan + cyclophosphamide | 1
  dexamethasone, then single-agent lenalidomide | 1
Best response prior to induction therapy [Number; unit: participants] — Best response was noted using the International Myeloma Working Group Guidelines: http://imwg.myeloma.org/international-myeloma-working-group-imwg-uniform-response-criteria-for-multiple-myeloma/
  participants
    Complete Response | 1
    partial Response | 27
    Stable Disease | 10

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Drug Combination as Therapy for Myeloma (Overall Response Rate)
Description: Myeloma response criteria developed by Bladé et al. was used to categorize response.
Time Frame: Best response at any point during each respective study phase was collected - once after consolidation/prior to mobilization (approximately 6 cycles after start of treatment), and once after mobilization
Population: All 38 patients were treated with DoVeD consolidation therapy (Vel + DEX with or without DOXIL). Of the 38 patients enrolled, 27 proceeded to mobilization (11 did not undergo mobilization). Responses were assessed prior to mobilization (post DoVED), and again after mobilization, to see if mobilization improved patient response.
Measure: Number; unit: participants
Groups:
- Treatment Arm - Post Mobilization: This is the response rate assessed for patients after their bortezomib-based mobilization.
- Treatment Arm - Responses Prior to Mobilization: This is the overall best response rate (ORR, ≥PR, as measured by ≥50% reduction in M-protein) to DoVeD therapy from post-primary induction (pre-DoVeD).
Arm/Group | Treatment Arm - Post Mobilization | Treatment Arm - Responses Prior to Mobilization
Number analyzed (Participants) | 27 | 38
participants
  Stringent Complete Response (sCR) | 4 | 0
  Complete Response (CR) | 3 | 1
  Very Good Partial response (VGPR) | 6 | 1
  Partial Response (PR) | 13 | 2
  Other Response (progression, stable disease, etc) | 1 | 6

2. Secondary Outcome: Yield of CD34+ Stem Cells
Description: This is the yield of CD34+ stem cells collection after high dose cyclophosphamide.
Time Frame: Occurred after mobilization, and prior to Stem cell transplant; a 7 day limit was imposed on stem cell collection
Measure: Median (Full Range); unit: 10^6 cells/kg
Groups:
- Treatment Arm - Post Bortezomib-based Mobilization: Yield of stem cell collection for the group that underwent bortezomib-based Mobilization
Arm/Group | Treatment Arm - Post Bortezomib-based Mobilization
Number analyzed (Participants) | 27
10^6 cells/kg | 23.2 [6.8 to 294.2]

3. Secondary Outcome: Progression Free Survival
Description: Response was assessed using IMWG guidelines, which for progressive disease are as follows:
  Increase of > 25% from lowest response value in any one or more of the following:
  * Serum M-component and/or (the absolute increase must be > 0.5 g/dL)*
  * Urine M-component and/or (the absolute increase must be > 200 mg/24 h)
  * Only in patients without measurable serum and urine M-protein levels; the difference between involved and uninvolved FLC levels. The absolute increase must be > 10 mg/dL
  * Bone marrow plasma cell percentage; the absolute percentage must be > 10%
  * Definite development of new bone lesions or soft tissue plasmacytomas or definite increase in the size of existing bone lesions or soft tissue plasmacytomas
  * Development of hypercalcaemia (corrected serum calcium > 11.5 mg/dL or 2.65 mmol/L) that can be attributed solely to the plasma cell proliferative disorder IF starting M protein component is > 5g/dL, then absolute increase of 1g is sufficient for progression.
Time Frame: Date of progression, assessed from start of trial to Final data cut off date (15 April 2011)
Measure: Median (Full Range); unit: months
Arm/Group | Treatment Arm (All Patients)
Number analyzed (Participants) | 38
months | 46.6 [6.4 to 68.8]

ADVERSE EVENTS:
Time Frame: Safety was monitored throughout the study, from start of study until when patients were removed (for either progression, toxicity, or to get a HD-SCT, which occurred up to 1 year after start of treatment).
Description: Safety was monitored throughout the study and adverse events (AEs) were graded by NCI-CTCAE version 3.0.
Arm/Group | Treatment Arm (All Patients)
Serious Adverse Events (participants affected / at risk) | 1/38
Other Adverse Events (participants affected / at risk) | 38/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Arm (All Patients) (N=38)
diarrhea (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Arm (All Patients) (N=38)
dizziness (General disorders) | 4 — DOVED consolidation phase
insomnia (Psychiatric disorders) | 22 — DOVED consolidation phase
depression (Psychiatric disorders) | 6 — DOVED consolidation phase
anxiety (Psychiatric disorders) | 5 — DOVED consolidation phase
irritability (Psychiatric disorders) | 3 — DOVED consolidation phase
nervousness (Psychiatric disorders) | 3 — DOVED consolidation phase
confusion (Psychiatric disorders) | 3 — DOVED consolidation phase
dry skin (Skin and subcutaneous tissue disorders) | 3 — DOVED consolidation phase
pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 — DOVED consolidation phase
cough (Respiratory, thoracic and mediastinal disorders) | 12 — DOVED consolidation phase
sinusitis (Respiratory, thoracic and mediastinal disorders) | 2 — DOVED consolidation phase
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 4 — DOVED consolidation phase
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 6 — DOVED consolidation phase
hearing impariment (Ear and labyrinth disorders) | 2 — DOVED consolidation phase
epistaxis (General disorders) | 3 — DOVED consolidation phase
sore throat (Ear and labyrinth disorders) | 2 — DOVED consolidation phase
blurred vision (Eye disorders) | 13 — DOVED consolidation phase
chest pain (Cardiac disorders) | 2 — DOVED consolidation phase
hypertension (Cardiac disorders) | 3 — DOVED consolidation phase
myopathy (Musculoskeletal and connective tissue disorders) | 5 — DOVED consolidation phase
pain in extremity (Musculoskeletal and connective tissue disorders) | 4 — DOVED consolidation phase
muscle weakness (Musculoskeletal and connective tissue disorders) | 7 — DOVED consolidation phase
cramping (Musculoskeletal and connective tissue disorders) | 2 — DOVED consolidation phase
back pain (Musculoskeletal and connective tissue disorders) | 7 — DOVED consolidation phase
weight gain (General disorders) | 3 — DOVED consolidation phase
fatigue (General disorders) | 24 — DOVED consolidation phase
dry mouth (General disorders) | 2 — DOVED consolidation phase
fever (General disorders) | 3 — DOVED consolidation phase
edema (Vascular disorders) | 13 — DOVED consolidation phase
headache (General disorders) | 6 — DOVED consolidation phase
taste alteration (General disorders) | 5 — DOVED consolidation phase
diarrhea (Gastrointestinal disorders) | 2 — mobilization phase
nausea (Gastrointestinal disorders) | 6 — mobilization phase
peripheral neuropathy (sensory) (Nervous system disorders) | 6 — mobilization phase
tremor (Nervous system disorders) | 2 — mobilization phase
insomnia (Psychiatric disorders) | 2 — mobilization phase
anxiety (Psychiatric disorders) | 3 — mobilization phase
cough (General disorders) | 3 — mobilization phase
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 2 — mobilization phase
fatigue (General disorders) | 7 — mobilization phase
fever (Infections and infestations) | 3 — mobilization phase
edema (Vascular disorders) | 2 — mobilization phase
headache (General disorders) | 2 — mobilization phase
thrombocytopenia (Blood and lymphatic system disorders) | 6 — DOVED consolidation phase
afebrile neutropenia (Blood and lymphatic system disorders) | 2 — DOVED consolidation phase
anemia (Blood and lymphatic system disorders) | 5 — DOVED consolidation phase
diarrhea (Gastrointestinal disorders) | 9 — DOVED consolidation phase
abdominal pain (Gastrointestinal disorders) | 6 — DOVED consolidation phase
dyspepsia (Gastrointestinal disorders) | 5 — DOVED consolidation phase
anorexia (Metabolism and nutrition disorders) | 2 — DOVED consolidation phase
constipation (Gastrointestinal disorders) | 15 — DOVED consolidation phase
nausea (Gastrointestinal disorders) | 5 — DOVED consolidation phase
increased appetite (Gastrointestinal disorders) | 2 — DOVED consolidation phase
bloating (Gastrointestinal disorders) | 3 — DOVED consolidation phase
peripheral neuropathy (sensory) (Nervous system disorders) | 28 — DOVED consolidation phase
hand and foot syndrome (Nervous system disorders) | 7 — DOVED consolidation phase
tremor (Nervous system disorders) | 10 — DOVED consolidation phase

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less